CLINICAL TRIAL: NCT07029191
Title: SYMPA-VEIN : Pilot Study Evaluating the ACCUVEIN Superficial Vein Visualization Device for the Detection of Alterations in the Autonomic Nervous System
Brief Title: Screening for Alterations in the Autonomic Nervous System
Acronym: SYMPA-VEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 49RC25_0164; 2025-A00899-40 (Other: ANSM)
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Dysautonomia; ACCUVEIN; Superficial Veins; Sympathetic Nervous System; Standing Test
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Progressive standing test (Experimental): Healthy subjects
  Interventions: Other: Progressive standing test

INTERVENTIONS:
Other: Progressive standing test — Progressive raising test in successive steps in a healthy subject

SUMMARY:
Dysautonomia is an alteration of the autonomic nervous system that manifests itself in different forms, some of which are very disabling. Dysautonomia accompanies many pathologies. Its importance in public health is illustrated by an incidence of 20-70% in diabetes. It affects between 400,000 and 1.4 million patients in the French diabetic population alone. Dysautonomia is mainly investigated through alterations in the cardiovascular system's reactivity to various maneuvers. It involves a methodology that evaluates the functionality of the sympathetic nervous system. This methodology is reserved for specialized laboratories, limiting access to diagnosis. Dysautonomia is therefore commonly overlooked for lack of a simple, effective diagnostic tool.

ACCUVEIN is an augmented-reality venipuncture device. It projects the network of superficial veins onto the patient's skin. Our aim is to show that ACCUVEIN is capable of objectivizing the venoconstriction caused by activation of the sympathetic system in a healthy subject, such as when moving to a standing position. If ACCUVEIN has this capability, it would then represent a simple and rapid diagnostic tool for objectifying a venoconstriction defect in patients with dysautonomia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 40
* Subject affiliated with or benefiting from a social security plan
* Subject having signed an informed consent form
* Subject without known chronic illness or long-term treatment (oral contraceptive authorized for women)
* Subject without symptoms of dysautonomia
* Subject with no history of cardiovascular disease
* No history of loss of consciousness
* Subjects without regular and excessive alcohol consumption according to the WHO
* Non-smoker, non-vapoteur
* No chronic pain

Exclusion Criteria:

* Known ECG abnormality
* Pregnant women, parturients and nursing mothers
* Person deprived of liberty by administrative or judicial decision
* Person under compulsory psychiatric care
* Adult subject to a legal protection measure
* Persons unable to express their consent
* Subject unable to understand study objectives or instructions
* Subject in a period of exclusion from another study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Progressive standing test | Day 1
  If the subject's resting ECG is normal, the experimental session then begins with a progressive uprighting test of the subject in increments starting at 0° (the horizontal position) then moving on to 15°, then 30°, then 45° and finally 70°, the maximum upright head-up position, i.e. a total of 5 increments). Progressive verticalization is performed on a verticalization table used in standard autonomic nervous system assessment procedures. Three thoracic electrocardiographic electrodes and the blood pressure measurement finger pad on the right middle finger are positioned, then the left upper limb is stripped and held at heart level by a suitable support throughout the experimental procedure. The subject then lies down on the examination table. Each level is maintained for 5 minutes. At the end of the last 70° stop, the examination table is returned to the horizontal position.

SECONDARY OUTCOMES:
Blood pressure recording | Day 1
  Recording of blood pressure by the Finapres Nova system begins after 5 minutes' rest in the supine position, to allow the body to adapt to this position. The standing test then begins.
Heart rate recording | Day 1
  Heart rate recording by the Finapres Nova system begins after 5 minutes' rest in the supine position, to allow the body to adapt to this position. The standing test then begins.
ACCUVEIN | Day 1
  A photograph of the forearm, with the superficial veins highlighted by the ACCUVEIN device, is taken during the last minute of each stage.
Breathing test | Day 1
  To confirm the absence of dysautonomia, two very short tests are performed. These tests involve asking the subject to breathe according to the experimenter's instructions (inflate lungs, deflate lungs), who then imposes a normal breathing rhythm of 12 cycles per minute for one minute. The subject is then asked to stand up on his own and maintain this posture for 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No